CLINICAL TRIAL: NCT05037968
Title: A Prospective, Randomized, Multi-center Study to Assess the Performance of MagnEtOs Flex Matrix Mixed With Local Autograft Compared to Trinity Elite Mixed With Local Autograft in Patients Undergoing up to Four-level Instrumented poSterolatEral Lumbar/Thoraco-lumbar Fusion (PLF)
Brief Title: MagnetOs Flex Matrix Compared to Trinity Elite Mixed With Local Autograft in Patients Undergoing up to Four-level Instrumented Posterolateral Fusion
Acronym: PRECISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Kuros BioSciences B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAG-523-002
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease; Spine Fusion; Leg Pain and/or Back Pain
Keywords: Degenerative Disc Disease; Spine Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Intra-patient control. Each patient serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MagnetOs Flex Matrix (Experimental): MagnetOs Flex Matrix use in instrumented posterolateral fusion, 5cc-10cc mixed with local autograft bone in a 1:1 ratio per spine level at the randomized assigned side
  Interventions: Device: MagnetOs Flex Matrix
- Trinity Elite (Active Comparator): Trinity Elite is a cryopreserved, viable cellular allograft containing cancellous bone and demineralized cortical bone designed for surgical use, applied per spine level at the contralateral side. Trinity Elite will be used as a bone graft extender (mixed with local autograft)
  Interventions: Device: Trinity Elite

INTERVENTIONS:
Device: MagnetOs Flex Matrix — Procedure: Instrumented Posterolateral Lumbar Fusion
  Arms: MagnetOs Flex Matrix
Device: Trinity Elite — Procedure: Instrumented Posterolateral Lumbar Fusion
  Arms: Trinity Elite

SUMMARY:
This is a phase IV post-marketing study for MagnetOs Flex Matrix. MagnetOs Flex Matrix is a synthetic bone graft extender product that is routinely used by surgeons as a treatment for patients with degenerative disc disease and undergoing spinal fusion surgery.

In this study, MagnetOs Flex Matrix will be used according to the latest U.S. Instructions For Use, specifically as a bone graft extender mixed with autograft in a 1:1 vol.% in the posterolateral spine.

Trinity Elite will also be used according to its latest IFU approved in the US. Specifically, this cellular based allograft is an allograft intended for the treatment of musculoskeletal defects.

DETAILED DESCRIPTION:
In this study, following a screening period of a maximum of 30 days, 100 patients will undergo up to four-level instrumented posterolateral fusion (PLF) procedure. Prior to surgery, each patient will be randomized to receive MagnetOs Flex Matrix on the assigned side of the spine and Trinity Elite on the other at the diseased levels. They will be followed up at discharge, Week 2, Week 6, Month 3, Month 6, and Month 12. The primary endpoint will be analyzed at Month 12.

In this study, MagnetOs Flex Matrix will be applied according to the latest Instructions for Use approved in the United States. Specifically, MagnetOs Flex Matrix will be used as a bone graft extender mixed with autograft in a 1:1 vol% in patients with leg pain, and/or back pain requiring up to four-level instrumented posterolateral spine fusion procedure. The fusion procedure (PLF) will be left to the surgeon's discretion.

Radiographs will be obtained at Screening, Week 2, Week 6, Month 3, Month 6 and Month 12. CT-scans will only be obtained at Month 6 and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read/be read, understand, and provide written informed consent and has signed the Investigational Review Board (IRB) approved informed consent.
* Male or female patient ≥ 18 years old.
* Patients with leg pain, and/or back pain requiring up to four-level instrumented posterolateral lumbar/thoraco-lumbar fusion (T11 - S1)
* Failed conservative treatment (physical therapy, bed rest, medications, spinal injections, manipulations, or transcutaneous electrical nerve stimulation) for a minimum period of 3 months prior to study enrollment.

Exclusion Criteria:

* Requires > four-level fusion or expected to need secondary intervention within one year following surgery.
* Had prior PLF fusion or attempted PLF fusion at the involved levels
* Had previous decompression at the involved levels.
* Women who are or intend to become pregnant within the next 12 months
* To treat conditions in which general bone grafting is not advisable.
* In conditions where the surgical site may be subjected to excessive impact or stresses, including those beyond the load strength of fixation hardware (e.g., defect site stabilization is not possible).
* In case of significant vascular impairment proximal to the graft site.
* In case of severe metabolic or systemic bone disorders (e.g., osteogenesis imperfecta or Paget's Disease) that affect bone or wound healing.
* In case of acute and chronic infections in the operated area (soft tissue infections; inflammation, bacterial bone diseases; osteomyelitis).
* When intraoperative soft tissue coverage is not planned or possible.
* Receiving treatment with medication interfering with calcium metabolism.
* Had leg pain, and/or back pain related to a benign or malignant tumor.
* Had history or presence of active malignancy.
* Has known substance abuse, psychiatric disorder, or condition which, in the opinion of the investigator, may influence the healing or ability to comply with protocol requirements.
* Is involved in active litigation relating to his/her spinal condition.
* Has participated in an investigational study within 30 days prior to surgery for study devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion by CT Scan | Month 12
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by CT-scan at Month 12. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes.

SECONDARY OUTCOMES:
Radiographic Fusion by Plain Radiographs | Month 6 and Month 12
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by plain radiographs.
Radiographic Fusion by CT Scan | Month 6
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by CT-scan at Month 6. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes.
Functional Outcome by Oswestry Disability Index | Screening, Week 2, Week 6, Month 3, Month 6, Month 12
  Functional outcome by the Oswestry Disability Index questionnaire. Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living. The lower the percentage the higher the patient's functionality. 0-20% minimal disability, 80-100% significant disability.
Back and Leg Pain by Visual Analog Pain Scale (VAS) | Screening, Week 2, Week 6, Month 3, Month 6, and Month 12
  Change in back and leg pain using Visual Analog Pain Scale score. The patient completed questionnaire is a unidimensional measure of pain intensity using a continuous scale comprised of a horizontal line 10 centimeters (100 mm) in length. The line is anchored by "no pain" (score of 0) and "worst imaginable pain". A higher score indicates greater pain intensity.
Neurologic Status by Physical Exam | Screening, Week 2, Week 6, Month 3, Month 6, and Month 12
  Change in neurologic status by examination to document stable, improved, or deficits in condition. Stable or improved findings for lower extremities, specifically reflexes, muscle strength, sensory, and straight leg raise.
Success Rate | Week 2, Week 6, Month 3, Month 6, and Month12
  Number of patients with secondary surgical interventions (SSI's) such as revisions, re-operations, removals, supplemental fixations, or any other procedure that adjusts or removes part of the original implant configuration with or without replacement of the components within 12 months of surgery.

OTHER OUTCOMES:
Safety Endpoint - number of patients with Adverse Events | Screening up to 12 Months post-op
  The number of patients with Adverse Events from Screening up to Month 12 after surgery.
Safety Endpoint - number of patients with Serious Adverse Events | Screening up to 12 Months post-op
  The number of patients with Serious Adverse Events from Screening up to Month 12 after surgery
Safety Endpoint - number of patients with Adverse Device Effects | 12 Months
  The number of patients with Adverse Device Effects from Screening up to Month 12 after surgery.
Safety Endpoint - number of patients with Device Related Complications | 12 Months
  The number of patients with any complications considered to device related with 12 months after surgery.
Health Economic - Duration of Surgery | 12 Months
  Duration of surgery in minutes.
Health Economic - Duration of Hospitalization | 12 Months
  Duration of hospital stay in days.
Health Economic - Return to Work | 12 Months
  Time to return to work in days.
Health Economic - Quality of Life | 12 Months
  Change in Quality of Life measurement using EuroQol-5D/5L scoring

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Health Research Institute, Columbia, Maryland
  - Michigan Orthopedic Surgeons, Bloomfield Hills, Michigan
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - Huntsman Spinal Clinic, Salt Lake City, Utah
  - Inova Healthcare, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No